CLINICAL TRIAL: NCT01579266
Title: Validating a New Writer's Cramp Scale
Brief Title: Validating a New Writer s Cramp Scale
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120104; 12-N-0104
Record Dates: First submitted 2012-04-14; First posted 2012-04-17 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2016-10-25

CONDITIONS: Dystonia
Keywords: Writer's Cramp; Focal Hand Dystonia; Writer Cramp; Dystonia
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- People with writer s cramp develop tightness in arm muscles and abnormal hand posture when writing, which makes writing difficult or impossible. At present, there is no suitable rating scale to measure the symptoms of or disability associated with writer s cramp. Researchers want to videotape people performing simple writing tasks. They will then compare the performance of people with writer s cramp on these tasks to those of people without writer s cramp. This information will help develop a rating scale to evaluate writer s cramp.

Objectives:

- To develop a new rating scale for writer s cramp.

Eligibility:

- Individuals at least 18 years of age who have writer s cramp.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have one outpatient study visit that will last about 3 hours.
* Participants will perform tasks related to writing, such as writing passages and drawing spirals and loops. They will be videotaped during these tasks. They will repeat some of the writing tasks three more times; on paper attached to a writing tablet, directly on the writing tablet, and on a computer tablet.
* The angles made by the joints will be measured at rest not while writing

healthy volunteers.

DETAILED DESCRIPTION:
Objective: Writer s cramp (WC) causes significant discomfort and disability to those afflicted by this condition. Studies on WC have been hampered by the lack of objective, validated rating scales. In this study, we will test and validate new instruments to rate WC; the WC impairment scale (WCIS) and a new disability scale (WCDS).We will also collect exploratory data about biomechanics of the hand.

Study population: The study population will consist of 20 subjects. Ten patients with WC and 10 age and handedness matched HVs will constitute the study population.

Design: 10 patients with WC and 10 age- and handedness-matched HV will be videotaped while writing. The WCIS scores will be given to each subject by four blinded raters (Drs. Mark Hallett, Barbara Karp, Katherine Alter, and Camilo Toro) based on the videos. The patients will complete the WCDS. In addition, each individual will be asked to repeat some basic elements of the scale while writing on the screen of a tablet PC, and on the surface of a detached digitizing tablet in order to generate high temporal and spatial resolution pen tip position samples for further numerical analyses and scoring. The biomechanics of the hand will be measured using a published scale.

Outcome measures: Using the WCIS, inter and intra-rater reliability, internal consistency (Cronbach s alpha) face validity, and reproducibility will be measured in addition to other secondary outcomes. The ease of use by the raters will be assessed for each subject. Reproducibility of writing on tablet, writing on paper placed on a writing tablet, and writing on a tablet PC will be assessed. Finally, biomechanics of the hands of patients with WC will be compared with those of the unaffected healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria for patients with WC and age and handedness-matched HVs:

  * Subjects must be at least 18 years of age.
  * Subjects must be willing to be videotaped while writing.
  * Subjects must have regular hand function with the ability to write without an assistive device

EXCLUSION CRITERIA:

* Patients with WC:

  * Botulinum toxin (BTX) administration within 3 months of participation.
  * Unable to provide consent.
  * Patients taking oral medications for WC including muscle relaxants or other centrally-active medications such as antidepressants which may enhance tremors.
  * Medical conditions that affect hand function, such as stroke, nerve entrapment, tremor, parkinsonism, chorea, ataxia affecting the dominant hand.
* HVs:

  * Unable to provide consent.
  * Healthy volunteers taking oral medications that may affect motor function such as muscle relaxants or centrally-active medications including medications for psychiatric conditions like antidepressants and antipsychotics.
  * Healthy volunteers with abnormal hand function including medical conditions that may influence hand function, e.g., strokes, nerve entrapments, tremor, parkinsonism, chorea, ataxia and psychiatric conditions (such as psychosis and depression) affecting the dominant hand.
  * Have history of hand surgery and or hand trauma.
  * Have abnormal findings on medical history and physical exam.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03-21; Study Completion 2016-10-25

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wissel J, Kabus C, Wenzel R, Klepsch S, Schwarz U, Nebe A, Schelosky L, Scholz U, Poewe W. Botulinum toxin in writer's cramp: objective response evaluation in 31 patients. J Neurol Neurosurg Psychiatry. 1996 Aug;61(2):172-5. doi: 10.1136/jnnp.61.2.172. PMID 8708685
- [Background] Pekmezovic T, Svetel M, Ivanovic N, Dragasevic N, Petrovic I, Tepavcevic DK, Kostic VS. Quality of life in patients with focal dystonia. Clin Neurol Neurosurg. 2009 Feb;111(2):161-4. doi: 10.1016/j.clineuro.2008.09.023. Epub 2008 Nov 7. PMID 18995953
- [Background] Burke RE, Fahn S, Marsden CD, Bressman SB, Moskowitz C, Friedman J. Validity and reliability of a rating scale for the primary torsion dystonias. Neurology. 1985 Jan;35(1):73-7. doi: 10.1212/wnl.35.1.73. PMID 3966004